CLINICAL TRIAL: NCT06198283
Title: Effects of Pressure Garments With and Without Low Level Laser Therapy on Hypertrophic Hand Scar in Children With Burn
Brief Title: Effects of Pressure Garments on Hypertrophic Hand Scar in Burn Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/RHS & AHS/23/0763
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Burns Laser
Keywords: Burn scar, Hypertrophy Scar; Pressure garment,; Low level laser,
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group will be treated by low level laser therapy with pressure garments
  Interventions: Other: Low Level LASER Therapy with Pressure Garment
- Group B (Active Comparator): This group will receive low level LASER therapy without pressure garment
  Interventions: Other: Low Level LASER Therapy without Pressure Garment

INTERVENTIONS:
Other: Low Level LASER Therapy with Pressure Garment — This group will be treated by low level laser therapy with pressure garment (8-10hrs a day) by Laplace' s Law method because it is more accurate since the range of pressures that can be delivered to a particular range of body circumferences varies depending on the fabric used and its particular tension- extension profile, the method is difficult to utilize manually and till present there is no available design tool to aid in its application. Pressure garments generate an increase in subdermal pressures in the range 9- 90 mmHg depending on the anatomical site. Garments over soft tissues generate pressures ranging from 9 to 33 mmHg. Over bony prominences the pressures range from 47 to 90 mmHg. 25mmHg pressure will be provided by garments and garments will be replaced in every 2 months
  Arms: Group A
Other: Low Level LASER Therapy without Pressure Garment — This group will receive low level LASER therapy (422-800nm) without pressure garment only for the duration of 6 weeks (3 days in a week with 20-30 minutes per session).
  Arms: Group B

SUMMARY:
Burns are type of injury that affect the skin or other tissues and are typically caused by acute trauma, including thermal sources, electricity, chemicals, friction, or radiation. Thermal burns are frequently caused by exposure to high temperature solids or liquids, as well as flames. The epidermis is the only layer of skin affected by superficial burns (sometimes known as "first degree" burns). Blistering is a common symptom of partial thickness (second degree) burns, which damage both the epidermis and dermis.

DETAILED DESCRIPTION:
This study will include patients with age 2-10 & having burns on hands and develop scars will be recruited through Randomized Controlled trial in which convenience sampling technique will be used. Two groups will be formed in which participants will be divided by lottery method. Group A which will be treated by low level laser therapy with pressure garment (8-10hrs a day) and group B which will receive low level LASER therapy (422-800nm) without pressure garment only for the duration of 6 weeks (3 days in a week with 20-30 minutes per session). Vancouver Scar Scale and PSOAS tool will be used. The result after statistical analysis will either show both treatments equally effective or not. Data will be calculated before and after treatment with the help of outcome measure tools. Results will be analyzed on SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-10 years
* Patient with 2nd degree of burns on hands and develop scar
* Patients after 3 months of burn on hand
* Only patients that were diagnosed with hypertrophic scars secondary to burn injuries were included
* Patients those with second degree burns or more or those with HS from burns
* Scar type (hypertrophic, flat or atrophic) and scar dyschromia (i.e. erythema) are the main factors that drive laser device selection

Exclusion Criteria:

* Participants who have certain medical problems that may impair scar healing or response to therapy interventions (such as uncontrolled diabetes, autoimmune disorders, or immunocompromised states).
* Those who have suffered burns recently (within the past few weeks) or who have had their scars for a long time (five years or more)
* Wounds that have open area and risk of bleeding occurs.
* Any spinal cord injuries.
* Patients with any other skin disease like skin cancer, inflammation,Allergic conditions etc
* Patients with under treatment like radiations etc

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Patient and observer Scar Assessment scale (POSAS) | 6 weeks
  The patient and observer scar evaluation scale (POSAS) was developed to objectively grade different scars based on the opinions of both the patient and an observer. The ease of use and comprehensive information it delivers make this instrument preferable to others. It was applied to the assessment of burn scars and linear surgical scars, with results that were both reliable and valid.Predictive validity was considered excellent with a AUC of 0.9, good from 0.8 to 0.899, adequate from 0.7 to 0.799 and poor when <0.7. A scale is considered internally consistent with a Cronbach' s alpha from0.70 to 0.90. For ICCs a minimum value of 0.70 was considered as an acceptable reliable result.
Vancouver Scar Scale VSS | 6 weeks
  The Vancouver Scar Scale (VSS), formerly called the Burn Scar Index, is the most used objective scar grading system. It was created in 1990. The VSS has a total score out of 13, broken down into four categories: pigmentation, vascularity, pliability, and scar height. The VSS isn't perfect because it doesn't take into account the patient's perspective, is subject to operator- dependent errors, leaves out discomfort and pruritis, and doesn't hold anyone responsible for huge scars with uneven coloration. Nonetheless, because of its intended use in assessing burn scars, it has become the most popular and widely-used scale of its kind.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Hammad Subhani, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noorbakhsh SI, Bonar EM, Polinski R, Amin MS. Educational Case: Burn Injury-Pathophysiology, Classification, and Treatment. Acad Pathol. 2021 Nov 28;8:23742895211057239. doi: 10.1177/23742895211057239. eCollection 2021 Jan-Dec. PMID 34869832
- [Background] Alnababtah K, Khan S, Ashford R. Socio-demographic factors and the prevalence of burns in children: an overview of the literature. Paediatr Int Child Health. 2016 Feb;36(1):45-51. doi: 10.1179/2046905514Y.0000000157. Epub 2014 Oct 13. PMID 25309999